CLINICAL TRIAL: NCT06604507
Title: Feasibility of Using an App for Managing Phantom Limb Pain Associated with Combat Amputation in Ukraine: a Quantitative & Qualitative Observational Trial in the 'Prevention and Management of Phantom Limb Pain' Project
Brief Title: Feasibility of Using an App for Managing Phantom Limb Pain Associated with Combat Injury in Ukraine (PAMELA)
Acronym: PAMELA
Status: Not yet recruiting | Type: Observational
Sponsor: Winfried Meißner (Other)
Responsible Party: Sponsor-Investigator, Winfried Meißner, Winfried Meissner, Jena University Hospital
Organization: Jena University Hospital (Other)
Other Study IDs: 2023-10-01
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Amputation, Traumatic; Pain, Phantom; Pain, Acute; Pain, Chronic; Pain, Neuropathic; Rehabilitation; War-Related Trauma
Keywords: Non-pharmacological treatment; App, computer; amputation, traumatic; pain, phantom; pain, acute; pain, chronic; pain, neuropathic; rehabilitation; war-related trauma
MeSH Terms: conditions — Amputation, Traumatic; Phantom Limb; Acute Pain; Chronic Pain; Neuralgia; War-Related Injuries; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Soldiers or civilians, who underwent an amputation as a result of the 2022 war in Ukraine: The cohort consists of soldiers or civilians, who underwent an amputation as a result of the 2022 war in Ukraine, and will use an app that provides non-pharmaceutical methods to care for the sensations and pains related to amputation.
  Interventions: Device: non-pharmacological app

INTERVENTIONS:
Device: non-pharmacological app — Amputees will be offered use of an app which offers a variety of non-pharmacological management techniques and exercises aimed at reducing the sensations and pain which are associated with amputation. These include: (1) offering information about the amputation, (2) augmented reality, this is a method for altering a person's perception about the real-world environment using computer simulation; (3) methods for reducing stress, also called 'Mindfulness-Based-Stress-Reduction' and (4) a method called 'Graded Motor Imagery' which aims to train the brain to address the changes which have occurred due to the amputation and which are related to pain and challenges with movement

SUMMARY:
In Ukraine, since the beginning of the full-scale war on February 24, 2022, a large number of individuals have lost a limb(s). Many of these amputees cannot access appropriate care in terms of pain management and rehabilitation. Consequently, healthcare providers in Ukraine have been seeking assistance from international, professional bodies to improve the care offered to amputees - soldiers and civilians.

Pain related to an amputation is chronic and so non-pharmacological approaches, rather than pharmacological, are appealing. In Germany, Routine Health, in Düsseldorf, have developed an app-based platform which offers amputees a variety of non-pharmacological management techniques.

In the PAMELA project, we will offer amputees and therapists in Ukraine, use of this app.

The app has been adapted for use in Ukraine.

The study will be carried out in 2 phases:

1. A pilot in 5 rehabilitation centers to assess feasibility of using the app during one pre-defined 8-week treatment cycle, tailored to each amputee; amputees will be offered to use the app for another 4 weeks, independently
2. Updating the app, based on experience gained in the pilot phase and sharing the app with amputees who wish to us it.

DETAILED DESCRIPTION:
In Ukraine, since the beginning of the full-scale war on February 24, 2022, approximately 50,000 individuals have lost a limb(s). Many of these amputees cannot access appropriate care in terms of pain management and rehabilitation. Consequently, healthcare providers in Ukraine have been seeking assistance from international, professional bodies to improve the care offered to amputees - soldiers and civilians.

The protocol outlined here is of a study which will offer amputees, and their therapists in Ukraine, support in treating pains associated with amputation, using non-pharmaceutical methods.

Pain related to an amputation is chronic and so non-pharmacological approaches, rather than pharmacological, are appealing. In Germany, Routine Health, in Düsseldorf, have developed an app-based platform which offers amputees a variety of non-pharmacological management techniques. In Germany, the app is s used by amputees injured in work-related accidents. The developers have gained extensive experience over the last 7 years in terms of the app's usability and its effect on amputation-related pains.

In the PAMELA project, we will offer amputees and therapists in Ukraine, use of this app. We anticipate that an app-based solution can be feasible as many of the amputees are young and, therefore, computer savvy, many as said to be motivated to regain their independence after their injury. With the limited resources in terms of availability healthcare professionals in Ukraine, we anticipate that offering amputees an app-based tool, which can be, used in different environments, hospital, rehabilitation centers or home, at different phases of their treatment, might be an effective and cost effective means for managing amputation-related pains.

The app has been adapted for use in Ukraine - modules have been translated into Ukrainian and we devised methodology for assessing demographics of the amputees, information about the injury and amputation-related pain and other symptoms. The literature stresses that when proving this form of non-pharmacological management, it is important to select suitable candidates, train them and tailor their care. Thus, at least for the first phase of the study (='pilot'), staff from Routine Health will train Ukrainian therapists (physiotherapists and occupational therapists) from 5 centers on how to use the app and they will recruit amputees in the center in which they work.

The study will be carried out in 2 phases:

1. A pilot in 5 rehabilitation centers to assess feasibility of using the app during one pre-defined 8-week treatment cycle, tailored to each amputee; amputees will be offered to use the app for another 4 weeks, independently
2. Updating the app, based on experience gained in the pilot phase and sharing the app with amputees who wish to us it.

ELIGIBILITY:
Inclusion Criteria:

* Amputee has given written informed consent for participation in the study.
* Male or Female
* Age - no restriction but adult
* Have undergone amputation of one limb, upper or lower.

Exclusion Criteria:

For Graded Motor Imagery / Mirror therapy Amputees with disorders such as post-traumatic stress disorders should perform mirror therapy only after initial assessment by the therapist carrying out the treatment, as the mirror image of two intact limbs might elicit memories associated with the trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People in Ukraine, soldiers or civilians, who have undergone an amputation of one limb, upper or lower, since the 2022 war.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of amputees completing a pre-defined 8-week Routine Health treatment protocol, tailored to each amputee. | 8 weeks
  To assess the feasibility of amputees cared for in rehabilitation centers in Ukraine being able to complete a pre-defined 8-week Routine Health treatment protocol, tailored to each amputee.
  This includes [i] whether the protocol was followed in terms of implementing the modules (duration & frequency) and [ii] whether the assessments of the amputation-related outcomes, at the different assessment time points, were filled in.

SECONDARY OUTCOMES:
Usability and acceptability of the app | 8 weeks after use of the app
  Assess usability and acceptability of the app by amputees & carers at 8 weeks.
Profile of amputees who completed the 8 week treatment protocol vs did not | 8 weeks after use of the app
  Assess the profile of patients who were able to complete the 8-week treatment protocol vs those who did not. Assess in terms of demographics, type of injury, character of pain
Pain-related amputation patient reported outcomes | Baseline, weekly for 12 weeks (8 weeks treatment with therapist, 4 weeks independent use)
  Assess information about pain-related patient reported outcomes obtained from the assessments carried out at baseline (=anamnesis), once weekly during the 8 week treatment and once weekly for another 4 weeks of independent use.
Profile of amputees who completed the 4 week independent use of the app vs did not | weeks 9 - 12 of app use
  Assess the profile of patients who wished to continue using the app, independently, for an additional 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Meissner, MD, Principal Investigator — Jena University Hospital; Volodymyr Romanenko, MD, Principal Investigator — Vita Medical
Locations (5):
- Ukraine (5):
  - University Clinic of Kharkiv National Medical University, Kharkiv
  - Kyiv Main Military Clinical Hospital, Kyiv
  - Odesa 10th City Hospital, Odesa
  - Vinnytsia National Medical University, Vinnytsia
  - Vinnytsia Prometei Pain Treatment Center, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during this study will be available for sharing with researchers. The data shared will include de-identified participant demographic information, longitudinal pain-related patient reported outcomes, information about the amputation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be available for sharing following publication of the study results and will remain accessible for up to 5 years.
Access Criteria: Data will be available upon reasonable request to researchers affiliated with academic, research, or healthcare institutions.
  Researchers interested in accessing the data will be required to submit a detailed research proposal outlining the intended use of the data.
  Sharing of the data will be contingent to approval from the study PIs and to researchers signing a data use agreement.
  People wishing to access data should write to:
  WINFRIED.Meissner@med.uni-jena.de
URL: https://pamela.in.ua

REFERENCES:
- [Background] Rothgangel A, Braun S, de Witte L, Beurskens A, Smeets R. Development of a Clinical Framework for Mirror Therapy in Patients with Phantom Limb Pain: An Evidence-based Practice Approach. Pain Pract. 2016 Apr;16(4):422-34. doi: 10.1111/papr.12301. Epub 2015 Apr 16. PMID 25880456
- [Background] Rothgangel A, Braun S, Smeets R, Beurskens A. Feasibility of a traditional and teletreatment approach to mirror therapy in patients with phantom limb pain: a process evaluation performed alongside a randomized controlled trial. Clin Rehabil. 2019 Oct;33(10):1649-1660. doi: 10.1177/0269215519846539. Epub 2019 May 8. PMID 31066315
- [Background] Kumar A, Soliman N, Gan Z, Cullinan P, Vollert J, Rice ASC, Kemp H. A systematic review of the prevalence of postamputation and chronic neuropathic pain associated with combat injury in military personnel. Pain. 2024 Apr 1;165(4):727-740. doi: 10.1097/j.pain.0000000000003094. Epub 2023 Dec 15. PMID 38112578
- See also: The website is intended for multidisciplinary healthcare providers, amputees and their families in Ukraine. It will offer information about surgery, pain management and rehabilitation of amputation, which an emphasis of traumatic amputation. — https://pamela.in.ua